CLINICAL TRIAL: NCT01650025
Title: Effects of the Probiotic Preparation VSL#3 on the Metabolic, Endocrine, Lipidomic and Inflammatory Parameters as Well as Variation of the Microbiota in Pediatric Patients With Body Mass Index >90°
Brief Title: Effects of VSL#3 on Metabolic, Endocrine, Lipidomic and Inflammatory Parameters of Pediatric Patients With BMI>90°
Acronym: VAIIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, Pediatrician, Hepatologist, Chief of Hepato-metabolic disease Unit Head of Liver Research Unit, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VAIIO
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: probiotic, obesity, BMI, metabolic profile, metabolomics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 placebo (Placebo Comparator): The placebo comparator is administered in the same form and dose as the active ingredient. The patient will take 2 sachets a day for 4 months.
  Interventions: Other: VSL#3 placebo
- VSL#3 active probiotic (Active Comparator): VSL#3 is a probiotic preparation containing 8 different strains of lactic acid bacteria and bifidobacteria. Each sachet contains 450 billion bacteria and the patient will be requested to take 2 sachets a day for 4 months
  Interventions: Dietary Supplement: VSL#3 active probiotic

INTERVENTIONS:
Dietary Supplement: VSL#3 active probiotic
  Other Names: VSL#3
  Arms: VSL#3 active probiotic
Other: VSL#3 placebo
  Other Names: placebo
  Arms: VSL#3 placebo

SUMMARY:
Obesity in children has become a significant social problem considering that nowadays 4 to 5 % of all children are obese in the industrialized countries with increased incidence in Europe by 10 to 50% over the past 10 years. Obesity is associated with the metabolic syndrome in 30% of the children and is considered as a state of chronic inflammation inducing the production of pro-inflammatory cytokines which determine metabolic and endocrine alterations on the organism. It has been observed that obesity is also linked to a change in the intestinal microflora with a reduction of Bacterioides and bifidobacteria and a decrease of Firmicutes and Staphylococcus aureus. The qualitative and quantitative analysis of the metabolites may provide us with a characterization of the existing phenotypes and variations in relation to the changes of the physiological state, in particular when supplemented or not with a probiotic preparation.

ELIGIBILITY:
Inclusion Criteria:

* age 6-12
* parents or tutors able to give the written consent and follow the study procedures Value of BMI>90°

Exclusion Criteria:

* - Any severe or concomitant clinical or psychiatric condition that, in the investigator's opinion, could affect the treatment, the evaluations and the inclusion in the protocol;
* Evidence of active liver disease due to other causes;
* Steroid treatment; immuno suppressive therapies, chemotherapy agents within 2 month from screening;
* Pregnancy or breastfeeding;
* Abuse of alcohol and drugs clinically relevant;
* Diabetes.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of VSL#3 on metabolic, endocrine, lipidomic, metabolomic and inflammatory markers and microbiota variation of pediatric patients with BMI>90° | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Nobili, PhD, Principal Investigator — Bambino Gesù Children Hospital
Locations (1):
- Bambino Gesù Children Hospital, Rome, Italy

REFERENCES:
- [Derived] Alisi A, Bedogni G, Baviera G, Giorgio V, Porro E, Paris C, Giammaria P, Reali L, Anania F, Nobili V. Randomised clinical trial: The beneficial effects of VSL#3 in obese children with non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2014 Jun;39(11):1276-85. doi: 10.1111/apt.12758. Epub 2014 Apr 16. PMID 24738701